CLINICAL TRIAL: NCT00523822
Title: Sacroiliac Orthopedic Blocking and Cervical Spine Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: RD0524070092
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Musculoskeletal Diseases
Keywords: This study seeks to determine if the correction of a sacroiliac lesion can produce a functional change in cervical spine.
MeSH Terms: conditions — Musculoskeletal Diseases

INTERVENTIONS:
Other: Spinal Manipulative Therapy

SUMMARY:
This study seeks to determine if the correction of a sacroiliac lesion can produce a functional change in cervical spine. Reduction of a sacroiliac joint lesion may alter cervical spine function.

ELIGIBILITY:
Inclusion Criteria:

* Young adults currently enrolled at Logan College

Exclusion Criteria:

* Recent cervical spine injuries or surgeries
* Surgical hardware in the cervical spine or pelvis
* Any cervical condition that would make ROM & strength testing painful.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kristan Giggey, DC, Principal Investigator — Logan College
Locations (1):
- Logan College, Chesterfield, Missouri, United States